CLINICAL TRIAL: NCT02977351
Title: Determining the Relationship Between the Atherosclerosis and Periodontopathogenic Microorganisms in Chronic Periodontitis Patients
Brief Title: Determining the Relationship Between the Atherosclerosis and Periodontopathogenic Microorganisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Dr. A. Seckin ERTUGRUL, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IzmirKCU
Record Dates: First submitted 2016-11-15; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerosis; Chronic Periodontitis
Keywords: Periodontopathogenic microorganisms; Non-surgical periodontal treatment
MeSH Terms: conditions — Atherosclerosis; Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atherosclerosis (Experimental): Patients with atherosclerosis and chronic periodontitis
  Interventions: Procedure: Non-surgical periodontal treatment
- Systemically healthy (Active Comparator): Patients with Systemically healthy and chronic periodontitis.
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment

SUMMARY:
Determine the relationship between the systemic indications of atherosclerosis by means of the change in the ratio of periodontopathogenic microorganisms following periodontal treatment of individuals who have been diagnosed with chronic periodontitis-atherosclerosis and for individuals who have been diagnosed with systemically healthy-chronic periodontitis.

DETAILED DESCRIPTION:
It has been aimed in this study to compare 1) the change in periodontal status; 2) the change of the periodontopathogen microorganisms (A. actinomycetemcomitans, P. gingivalis, T. forsythia, T. denticola, P. intermedia, P. micros, F. nucleatum/periodonticum, C. rectus, E. nodatum, E. corrodens, and C. gingivalis/ochracea/sputigena) in dental plaque samples, 3) the changes of the amounts of HDL, LDL, hs-CRP white blood cell levels (WBC), platelet levels (PLT), creatinine, and fibrinogen in serum samples; and 4) the correlation between periodontopathogen microorganisms (A. actinomycetemcomitans, P. gingivalis, T. forsythia, T. denticola, P. intermedia, P. micros, F. nucleatum/periodonticum, C. rectus, E. nodatum, E. corrodens, and C. gingivalis/ochracea/sputigena) and HDL, LDL, hs-CRP WBC, PLT, creatinine, and fibrinogen in patients that have been diagnosed with atherosclerosis-chronic periodontitis and systemic healthy patients and patients diagnosed with chronic periodontitis, following non surgical periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

* had no systemic disease,
* had not used any antibiotics
* had not used medications with an impact on the immune system,
* had not received any periodontal and/or medical treatment within the last 6 months.

Exclusion Criteria:

* smokers of cigarettes or other tobacco products,
* pregnant or breastfeeding,
* non-stable cardiovascular condition.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Periodontopathogenic microorganism levels | 1 year

IPD SHARING:
Plan to Share IPD: No